CLINICAL TRIAL: NCT02660385
Title: Cognitive Behavioral Therapy for Insomnia: A Self-Management Strategy for Chronic Illness in Heart Failure
Brief Title: Insomnia Self-Management in Heart Failure
Acronym: HSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Milton S. Hershey Medical Center (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0904005041a; R01NR016191 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Failure; Heart Failure; Congestive Heart Failure; Heart Failure, Congestive; Sleep Initiation and Maintenance Disorders; Chronic Insomnia; Disorders of Initiating and Maintaining Sleep; Fatigue; Pain; Depressive Symptoms; Sleep Disorders; Anxiety
Keywords: pain; insomnia; cardiac failure; sleep; fatigue; heart disease; anxiety; actigraphy; psychomotor vigilance; six minute walk; depression; cognitive behavioral therapy; self-management; self-care
MeSH Terms: conditions — Heart Failure; Sleep Initiation and Maintenance Disorders; Fatigue; Pain; Depression; Sleep Wake Disorders; Anxiety Disorders; Heart Diseases | interventions — Cognitive Behavioral Therapy; Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive behavioral therapy for insomnia (CBT-I) will be provided in a group format, led by an interventionist. CBT-I includes strategies for modifying thoughts and behaviors about sleep. Participants will be instructed on and practice methods for modifying their thoughts and behaviors about sleep and insomnia. Participants will participate in four sessions, conducted every other week for 8 weeks. They will receive a call from the interventionist on intervening weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Heart Failure Self-Management Education (Active Comparator): Heart Failure Self-management education is an intervention that will be provided by a nurse in a group format. This includes standard components, such as education about fluid and sodium management, heart failure medications, diet and physical activity. Participants will participate in four sessions, conducted every other week for 8 weeks. They will receive a call from the interventionist on intervening weeks.
  Interventions: Behavioral: Self-Management Education for Heart Failure

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — This behavioral intervention includes strategies for modifying thoughts, cognitions and behaviors regarding sleep provided by a therapist in a group format.
  Other Names: Self-management for insomnia
  Arms: Cognitive Behavioral Therapy
Behavioral: Self-Management Education for Heart Failure — This is an educational education designed to teach patients about self-management their heart failure. It includes information on medications, lifestyle, cardiac devices, diet, and when to seek assistance from a health care provider.
  Arms: Heart Failure Self-Management Education

SUMMARY:
Chronic insomnia may contribute to the development and exacerbation of heart failure (HF), incident mortality and contributes to common and disabling symptoms (fatigue, dyspnea, anxiety, depression, excessive daytime sleepiness, and pain) and decrements in objective and subjective functional performance.

The purposes of the study are to evaluate the sustained effects of CBT-I on insomnia severity, sleep characteristics, daytime symptoms, and functional performance over twelve months among patients who have stable chronic HF and chronic insomnia. The effects of the treatment on outcomes of HF (hospitalization, death) and costs of the treatment will also be examined.

A total of 200 participants will be randomized to 4 bi-weekly group sessions of cognitive behavioral therapy for CBT-I (behavioral was to improve insomnia and sleep) or HF self-management education.

Participants will complete wrist actigraph (wrist-watch like accelerometer) measures of sleep, diaries, reaction time, and 6 minute walk test distance. They will also complete self-report measures of insomnia, sleep, symptoms, and functional performance. In addition the effects on symptoms and function over a period of one year.

DETAILED DESCRIPTION:
Almost 75% of HF patients, a group of about 5.1 million Americans who have poor function and high levels of morbidity and mortality, report poor sleep. As many as 25-56% of HF patients report chronic insomnia (difficulty initiating or maintaining sleep or waking early in the morning, with non-restorative sleep that persists for at least a month). Chronic insomnia may contribute to the development and exacerbation of HF and incident mortality. It is also associated with common and disabling symptoms (fatigue, dyspnea, anxiety, depression, excessive daytime sleepiness, and pain) and decrements in objective and subjective functional performance.However, insomnia is under-diagnosed and under-treated in this population.

Cognitive behavioral therapy for insomnia (CBT-I) is a multi-modal behavioral treatment focused on modifying beliefs and attitudes about sleep and is efficacious in many populations. The purposes of RCT are to evaluate the sustained effects of CBT-I, compared with HF self-management education (attention control), on insomnia severity, sleep characteristics, daytime symptoms, and functional performance over twelve months among patients who have stable chronic HF and chronic insomnia and receive evidence-based HF disease management. We will also evaluate the cost-effectiveness of CBT-I compared with the attention-control condition and explore the effects of CBT-I on event-free survival. We will address the following specific aims (*primary outcomes): (1) Test the sustained effects (baseline - 2 weeks, 6, 9, 12 months) of CBT-I provided in 4 group sessions over 8 weeks, compared with HF self-management education (attention control condition), on: (1a) *insomnia severity and self-reported and actigraph-recorded sleep characteristics (*sleep quality, *sleep efficiency, sleep latency, and duration); (1b) symptoms (*fatigue, anxiety, depression, pain, sleepiness, sleep-related impairment), and psychomotor vigilance (PVT); and (1c) symptom clusters [membership in clusters characterized by severity of specific symptoms; transition between clusters over time]; (2) Test the sustained effects of CBT-I on self-reported and objective functional performance; and (3) Examine the cost-effectiveness of CBT-I. Exploratory aim: We will explore the effects of CBT-I on event-free survival.

A total of 200 patients will be randomized to 4 bi-weekly sessions of group CBT-I or an attention control condition consisting of HF self-management education. Wrist actigraph measures of sleep, diaries, psychomotor vigilance and 6 minute walk test distance, and self-report measures of insomnia, sleep, symptoms, and functional performance will be obtained at baseline and follow-up. Data analysis will consist of mixed effects models, latent transition analysis, stochastic cost-effectiveness analysis, and survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic heart failure, chronic insomnia, English speaking/reading,

Exclusion Criteria:

* untreated sleep disordered breathing or restless legs syndrome, rotating/night shift work, active illicit drug use, bipolar disorder, neuromuscular conditions affecting the non-dominant arm end-stage renal failure, significant cognitive impairment, unstable medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy S Redeker, PhD, Principal Investigator — Yale University School of Nursing
Locations (1):
- Yale University School of Nursing, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data collected for the primary study aims (participant demographics, clinical characteristics, treatment group assignment and primary study outcomes (insomnia severity, sleep quality, actigraph-recorded sleep characteristics), daytime symptoms, and functional performance. We will also make the health care utilization/cost data available.
Supporting Information: Study Protocol
Time Frame: The data will be made available starting in January 2025
Access Criteria: Access to the data can be requested through contact with the principal investigators, Nancy S. Redeker, PhD, RN, FAHA, FAAN Nancy.redeker@yale.edu

REFERENCES:
- [Derived] O'Connell M, Feder SL, Nwanaji-Enwerem U, Redeker NS. Focus Group Study of Heart Failure Nurses' Perceptions of the Feasibility of Cognitive Behavioral Therapy for Insomnia. Nurs Res. 2024 Mar-Apr 01;73(2):109-117. doi: 10.1097/NNR.0000000000000706. Epub 2023 Nov 9. PMID 37967228
- [Derived] Jeon S, Conley S, Hollenbeak C, O'Connell M, Wang Z, Tocchi C, Redeker NS. Rest-activity rhythms predict time to hospitalizations and emergency department visits among participants in a randomized control of adults with heart failure and insomnia. Sleep Med. 2023 Aug;108:1-7. doi: 10.1016/j.sleep.2023.05.019. Epub 2023 May 27. PMID 37301192
- [Derived] Redeker NS, Conley S, O'Connell M, Geer JH, Yaggi H, Jeon S. Sleep-related predictors of cognition among adults with chronic insomnia and heart failure enrolled in a randomized controlled trial of cognitive behavioral therapy for insomnia. J Clin Sleep Med. 2023 Jun 1;19(6):1073-1081. doi: 10.5664/jcsm.10498. PMID 36740924
- [Derived] O'Connell M, DeSanto Iennaco J, Linsky S, Jeon S, Conley S, Gaiser E 3rd, Redeker NS. Treatment Fidelity in a Randomized Controlled Trial of Cognitive Behavioral Therapy for Insomnia in Heart Failure. Nurs Res. 2022 Nov-Dec 01;71(6):459-468. doi: 10.1097/NNR.0000000000000616. Epub 2022 Aug 20. PMID 35997691
- [Derived] O'Connell M, Jeon S, Conley S, Linsky S, Redeker NS. Coping, symptoms, and insomnia among people with heart failure during the COVID-19 pandemic. Eur J Cardiovasc Nurs. 2023 Apr 12;22(3):291-298. doi: 10.1093/eurjcn/zvac072. PMID 35938348
- [Derived] Breazeale S, Jeon S, Hwang Y, O'Connell M, Nwanaji-Enwerem U, Linsky S, Yaggi HK, Jacoby DL, Conley S, Redeker NS. Sleep Characteristics, Mood, Somatic Symptoms, and Self-Care Among People With Heart Failure and Insomnia. Nurs Res. 2022 May-Jun 01;71(3):189-199. doi: 10.1097/NNR.0000000000000585. PMID 35149627
- [Derived] Redeker NS, Yaggi HK, Jacoby D, Hollenbeak CS, Breazeale S, Conley S, Hwang Y, Iennaco J, Linsky S, Nwanaji-Enwerem U, O'Connell M, Jeon S. Cognitive behavioral therapy for insomnia has sustained effects on insomnia, fatigue, and function among people with chronic heart failure and insomnia: the HeartSleep Study. Sleep. 2022 Jan 11;45(1):zsab252. doi: 10.1093/sleep/zsab252. PMID 34657160
- [Derived] Redeker NS, Knies AK, Hollenbeak C, Klar Yaggi H, Cline J, Andrews L, Jacoby D, Sullivan A, O'Connell M, Iennaco J, Finoia L, Jeon S. Cognitive behavioral therapy for insomnia in stable heart failure: Protocol for a randomized controlled trial. Contemp Clin Trials. 2017 Apr;55:16-23. doi: 10.1016/j.cct.2017.01.009. Epub 2017 Jan 31. PMID 28159703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used multiple recruitment strategies including clinic-based recruitment, letters to patients identified from electronic databases, the patient portal, brochures and posters placed in clinics, presentations to heart failure support groups, and online advertising
Pre-assignment Details: 195 enrolled. Six participants dropped out prior to randomization, and 189 were randomized to HH and HS conditions. Fourteen completed the intervention or control condition but dropped out or died before follow-up assessments began. 175 completed at least one follow-up assessment.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Started | 100 | 89
Completed | 91 | 84
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Population: We completed baseline analyses on 175 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education | Total
Number analyzed (Participants) | 91 | 84 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row total does not differ from Overall
  years | 62.0 (13.1) | 64.1 (12.6) | 63.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 53 | 47 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 86 | 80 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 69 | 64 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity
Description: Insomnia severity will be measured with the Insomnia Severity Index, a brief self-report instrument measuring patients' perception of their insomnia. The instrument includes 7 items assessing the severity of sleep onset and sleep maintenance difficulties, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a 0-4 scale (4 indicates greater severity) with a total score ranging from 0 to 28. Scores are categorized as not clinically significant, sub-threshold insomnia, moderate insomnia or severe insomnia.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale | -6.60 (5.23) | -3.46 (5.18)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0002, Generalized Linear Mixed Model (GLMM); GLMM with random intercepts and unstructured covariances with changes within groups and time-group interactions to compare the intervention effects; Effect Size = -0.60

2. Primary Outcome: Change in Fatigue
Description: The symptom of fatigue was measured with the PROMIS Item Bank v1.0 - Fatigue - Short Form 8a. The instrument measures a range of symptoms of fatigue from mild tiredness to exhaustion that may interfere with the performance of daily activities. The instrument uses a 7-day time frame and a 5-point rating scale that ranges from 1 ("Not at all") to 5 ("Very much"). The measure uses a T-score metric in which 50 is the mean of a relevant reference population (the general population) and 10 is the standard deviation (SD) of the population. Higher scores mean more fatigue. To find the total raw score we summed the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. We used the score conversion table to translate the total raw score into a T-score for each participant. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe. The range of scores is 33-78.
Time Frame: Baseline to 3 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score | -3.24 (3.16) | -1.13 (8.05)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0723, GLMM — GLMM with random intercepts and unstructured covariances with changes within groups and time-group interactions to compare the intervention effects

3. Primary Outcome: Change in Sleep Efficiency-measured With PSQI
Description: Sleep efficiency refers the ratio of time spent asleep to the amount of time spent in bed. Sleep efficiency will be subjectively measured with the Pittsburgh Sleep Quality Index, an instrument used to calculate self-reported sleep duration, sleep efficiency sleep latency, sleep disturbances, and global sleep quality. Items 1 (bed time), 3 (wake time) are used to determine time-in-bed (the difference between Q1 and Q3). Q4 is time asleep while in bed. Sleep efficiency= (time asleep/time in bed) * 100
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
percent | 4.87 (17.41) | -1.96 (15.41)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0110, GLMM; [statistical method as in outcome 1, analysis 1]; effect size = 0.42

4. Primary Outcome: Change in Sleep Quality
Description: Sleep Quality was subjectively measured with the Pittsburgh Sleep Quality Index, an instrument used to calculate self-reported sleep duration, sleep efficiency sleep latency, sleep disturbances, and global sleep quality. The 19 self-rated items are calculated to provide a global score of sleep quality ranging from 0-21, with "0" indicating no difficulty, and "21" indicating severe difficulty in all areas.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale | -2.78 (3.16) | -0.51 (3.31)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p < 0.0001, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.70

5. Primary Outcome: Change in Sleep Efficiency-measured With Actigraphy
Description: Sleep efficiency refers the ratio of time spent asleep to the amount of time spent in bed. Sleep efficiency was objectively measured using actigraphy, a method of inferring sleep from the presence or absence of wrist movement. Participants wore the Respironics Minimitter Actiwatch AW2, a wrist-worn actigraph, to elicit objective sleep efficiency for a two week period. Participants also completed a daily diary (lights out/on, times/purpose of removal, hypnotic use) for use in interpretation of actigraphy data.
  Sleep efficiency=(time asleep/time in bed) * 100
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
percent | -0.5 (5.8) | 0.3 (7.2)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.4356, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.12

6. Primary Outcome: Change From Baseline in Fatigue
Description: as for outcome 2
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score
  6 month change | -3.16 (0.70) | -1.37 (0.72)
  12 month change | -4.26 (0.67) | -1.49 (0.72)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0148, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

7. Primary Outcome: Change From Baseline in Insomnia Severity
Description: Insomnia severity will be measured with the Insomnia Severity Index, a brief self-report instrument measuring patients' perception of their insomnia. The instrument includes 7 items assessing the severity of sleep onset and sleep maintenance difficulties, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a 0-4 scale (4 indicates greater severity) with a total score ranging from 0 to 28. Scores are categorized as not clinically significant, sub-threshold insomnia, moderate insomnia or severe insomnia.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale
  6 month change | -6.63 (0.48) | -4.06 (0.49)
  12 month change | -6.69 (0.47) | -4.57 (0.50)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0130, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

8. Primary Outcome: Change From Baseline in Sleep Quality
Description: Sleep Quality was subjectively measured with the Pittsburgh Sleep Quality Index, an instrument used to calculate self-reported sleep duration, sleep efficiency sleep latency, sleep disturbances, and global sleep quality. The 19 self-rated items are calculated to provide a global score ranging from 0-21, with "0" indicating no difficulty, and "21" indicating severe difficulty in all areas.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale
  6 month change | -3.02 (0.31) | -0.92 (0.32)
  12 month change | -2.89 (0.32) | -1.36 (0.34)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0130, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

9. Primary Outcome: Change From Baseline in Sleep Efficiency Measured With PSQI (%)
Description: Sleep efficiency refers the ratio of time spent asleep to the amount of time spent in bed. Sleep efficiency will be subjectively measured with the Pittsburgh Sleep Quality Index, an instrument used to calculate self-reported sleep duration, sleep efficiency sleep latency, sleep disturbances, and global sleep quality. Items 1 (bed time), 3 (wake time) are used to determine time-in-bed (the difference between Q1 and Q3). Q4 is time asleep while in bed. Sleep efficiency= (time asleep/time in bed) * 100
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months to 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
percent
  6 month change | 5.21 (1.51) | 0.91 (1.52)
  12 month change | 4.91 (1.43) | 1.17 (1.49)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0130, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

10. Primary Outcome: Change From Baseline in Sleep Efficiency Measured With Actigraphy
Description: Sleep efficiency refers the ratio of time spent asleep to the amount of time spent in bed. Sleep efficiency was objectively measured using actigraphy, a method of inferring sleep from the presence or absence of wrist movement. Participants wore the Respironics Minimitter Actiwatch AW2, a wrist-worn actigraph, to elicit objective sleep efficiency for a two week period. Participants also completed a daily diary (lights out/on, times/purpose of removal, hypnotic use) for use in interpretation of actigraphy data. Sleep efficiency=(time asleep/time in bed) * 100
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
percent
  6 month change | -0.53 (0.51) | 0.17 (0.57)
  12 month change | -0.44 (0.58) | 0.01 (0.59)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.6358, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

11. Secondary Outcome: Change in Sleep Duration
Description: Sleep duration was objectively measured using actigraphy, a method of inferring sleep from the presence or absence of wrist movement. Participants will wear the Respironics Minimitter Actiwatch AW2, a wrist-worn actigraph, to elicit objective sleep duration for a two week period. Participants will also complete a daily diary (lights out/on, times/purpose of removal, hypnotic use) for use in interpretation of actigraphy data.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
hours | 0.24 (1.73) | -0.44 (2.11)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0318, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.35

12. Secondary Outcome: Change From Baseline in Sleep Duration
Description: Sleep duration was objectively measured using actigraphy, a method of inferring sleep from the presence or absence of wrist movement. Participants wore the Respironics Minimitter Actiwatch AW2, a wrist-worn actigraph, to elicit objective sleep duration for a two week period. Participants completed a daily diary (lights out/on, times/purpose of removal, hypnotic use) for use in interpretation of actigraphy data.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
hours
  6 month change | 0.21 (0.12) | -0.18 (0.12)
  12 month change | 0.03 (0.11) | -0.18 (0.12)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.2722, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

13. Secondary Outcome: Change in Anxiety Symptoms
Description: Anxiety symptoms were measured with the PROMIS - Anxiety V1.- Short Form 8a. The instrument measures fear (worry, panic), anxious misery (e.g., dread), hyperarousal (e.g., tension, restlessness), and somatic symptoms (e.g., dizziness). The instrument uses a 7-day time frame and a 5-point rating scale that ranges from 1 ("Never") to 5 ("Always"). The measure uses a T-score metric in which 50 is the mean of a relevant reference population (the general population) and 10 is the standard deviation (SD) of the population. Higher scores mean more anxiety symptoms. To find the total raw score we summed the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. We used the score conversion table to translate the total raw score into a T-score for each participant. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe. The range of scores is 37-84.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score | -2.08 (5.98) | -0.32 (7.16)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0954, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.27

14. Secondary Outcome: Change From Baseline in Anxiety Symptoms
Description: as for outcome 13
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score
  6 month change | -2.73 (0.73) | -1.67 (0.74)
  12 month change | -2.85 (0.71) | -1.90 (0.74)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.4222, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

15. Secondary Outcome: Change in Depressive Symptoms
Description: Depressive symptoms were measured with the PROMIS - Depression V1.- Short Form 8a. The instrument measures negative mood (sadness), views of self (worthlessness), and social cognition (loneliness), and decreased positive affect and engagement. The instrument uses a 7-day time frame and a 5-point rating scale that ranges from 1 ("Never") to 5 ("Always"). The measure uses a T-score metric in which 50 is the mean of a relevant reference population (the general population) and 10 is the standard deviation (SD) of the population. Higher scores mean more depressive symptoms. To find the total raw score we summed the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. We used the score conversion table to translate the total raw score into a T-score for each participant. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe. The range of scores is 38-82.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score | -1.93 (6.83) | -2.50 (6.37)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.5781, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.09

16. Secondary Outcome: Change From Baseline in Depressive Symptoms
Description: as for outcome 15
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score
  6 month change | -1.55 (0.66) | -2.549 (0.68)
  12 month change | -1.11 (0.64) | -2.71 (0.68)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.1238, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

17. Secondary Outcome: Change in Sleepiness
Description: Sleepiness was measured using the Epworth Sleepiness Scale (ESS). The ESS is an 8-item self report instrument used to measure general levels of daytime sleepiness or sleep propensity in adults. The instrument asks subjects to rate on a scale of 0 to 3 the chances that he or she would doze in each of eight different situations. ESS scores can range from 0 to 24, with higher scores indicating higher levels of daytime sleepiness.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale | -1.39 (4.21) | -0.23 (3.37)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0558, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.30

18. Secondary Outcome: Change From Baseline in Sleepiness
Description: Sleepiness will be measured using the Epworth Sleepiness Scale (ESS). The ESS is an 8-item self report instrument used to measure general levels of daytime sleepiness or sleep propensity in adults. The instrument asks subjects to rate on a scale of 0 to 3 the chances that he or she would doze in each of eight different situations. ESS scores can range from 0 to 24, with higher scores indicating higher levels of daytime sleepiness.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 6 and 12 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 6 months and 12 months
Population: Modified intention to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale
  6 month change | -1.99 (0.37) | -0.68 (0.37)
  12 month change | -2.15 (0.35) | -0.84 (0.36)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0230, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

19. Secondary Outcome: Change in Dyspnea
Description: Symptoms of dyspnea were measured with the Multidimensional Assessment of Dyspnea Scale, a 16-item instrument to measure self-reported shortness of breath and the effect of shortness of breath on daily activities. The items are used to calculate a global dyspnea index, with higher scores indicating more severe dyspnea and greater impact on activities of daily living. The range of possible scores are between 4 and 50. To calculate the Global Dyspnea Index (GDI), we converted item 15 to a 0 - 10 scale by multiplying each score by 2.5 and then finding the sum of items 1, 2, and 3, and average 4 - 14. We did not assign a score to items 4 - 14 if the respondent gave a response of "do not do activity." If a respondent selected "no shortness of breath" on item 1, we assigned a zero to items 2 - 16. Item 16 is not included in the GDI.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale | -0.77 (8.5) | 0.34 (8.3)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.4597, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.06

20. Secondary Outcome: Change From Baseline in Dyspnea
Description: as for outcome 19
Time Frame: Baseline to 6 months and 12 months
Population: Modified intent to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale
  6 month change | -0.12 (0.95) | 1.20 (0.94)
  12 month change | -1.32 (0.93) | 0.41 (0.95)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.1943, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

21. Secondary Outcome: Change in Psychomotor Vigilance
Description: Psychomotor vigilance will be measured with the Psychomotor Vigilance Test (PVT), a widely used measure of behavioral alertness that is highly sensitive to changes related to sleep deprivation. The 10-minute PVT measures sustained or vigilant attention by recording response times to visual (or auditory) stimuli that occur at random inter-stimulus intervals. Scoring includes a numerical measure of sleepiness by counting the number of lapses in attention of the tested subject.
Time Frame: Baseline to 3 months
Population: Modified intent to treat
Measure: Mean (Standard Deviation); unit: number of lapses
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
number of lapses | -0.10 (0.87) | -0.30 (0.98)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0027, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.23

22. Secondary Outcome: Change From Baseline in Psychomotor Vigilance
Description: as for outcome 21
Time Frame: Baseline to 6 months and 12 months
Population: modified intent to treat
Measure: Least Squares Mean (Standard Error); unit: number of lapses
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
number of lapses
  6 month change | -0.16 (0.09) | -0.55 (0.09)
  12 month change | -0.25 (0.09) | -0.48 (0.09)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0792, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

23. Secondary Outcome: Change in Functional Performance
Description: Functional performance was measured with the Medical Outcomes Study (MOS) SF36v2 Physical Functioning Scale. The SF36v2 is a multi-purpose self-reported health survey that yields an 8-scale profile of functional health and well-being. The physical functioning scale assesses performance of daily activities, with the lowest score indicating an individual who is very limited in performing all physical activities, including bathing or dressing, and the highest score indicating an individual who can perform all types of vigorous physical activity without limitations due to health. Physical functioning scores were calculated using the Quality Metric Outcomes TM Scoring Software 4.5, which uses norm-based scoring. The range of possible scores is from 0-100; the typical range of norm based physical functioning is 20 to 60.
Time Frame: Baseline to 3 months
Population: Modified Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale | -0.79 (13.5) | 1.17 (13.4)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0656, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.13

24. Secondary Outcome: Change From Baseline in Functional Performance
Description: as for outcome 23
Time Frame: Baseline to 6 months and 12 months
Population: Modified intent to treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
score on a scale
  6 month change | -0.61 (1.36) | 1.40 (1.40)
  12 month change | 0.06 (1.40) | 2.56 (1.46)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.2174, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

25. Secondary Outcome: Change in Distance (Feet) Traveled During Six Minute Walk Test
Description: Functional capacity was objectively measured using the Six Minute Walk Test, which measures the distance that an individual can quickly walk on a flat, hard surface in a period of 6 minutes. The test is self-paced, and evaluates the global and integrated responses of all physiological systems involved during exercise. Participants choose their own intensity of exercise and are allowed to stop and rest during the test. Results are reported as an absolute value (distance walked), and interpreted according to change in functional capacity over time.
  For clarification, when results were entered, the outcome measure title was edited to include "change in" and the time frame was changed to Baseline to 3 months. When registered, the original time frame did not accurately portray the amount of time in which follow up data were collected.
Time Frame: Baseline to 3 months
Population: Modified intention to treat
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
Feet | 74.7 (236.2) | 61.6 (156.3)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.7028, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.07

26. Secondary Outcome: Change in Distance (Feet) Traveled During Six Minute Walk Test
Description: Functional capacity was objectively measured using the Six Minute Walk Test, which measures the distance that an individual can quickly walk on a flat, hard surface in a period of 6 minutes. The test is self-paced, and evaluates the global and integrated responses of all physiological systems involved during exercise. Participants choose their own intensity of exercise and are allowed to stop and rest during the test. Results are reported as an absolute value (distance walked), and interpreted according to change in functional capacity over time.
Time Frame: Baseline to 6 months and 12 months
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: feet
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
feet
  6 month change | 101.0 (17.0) | 44.0 (16.6)
  12 month change | 117.4 (18.1) | 61.3 (17.7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0509, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

27. Secondary Outcome: Cost Effectiveness
Description: Cost effectiveness was evaluated in terms of direct costs for health care resources used (ED visits, hospitalizations, inpatient and outpatient visits), as well as indirect costs (time missed from work, travel, and self-management and CBT-I activities). Out-of-pocket expenses were estimated using self-reported medical history health care resource use data (e.g., visits to health care providers, hospitalizations, emergency department visits). Information on costs were obtained by self-report and validated through the EMR, hospital cost accounting database, and the Medicare fee schedule.
Time Frame: 12 months post treatment
Population: Participants in trial who had complete self-reported indirect cost data.
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 79 | 71
dollars
  Cardiology visits | 32 [16 to 48] | 42 [18 to 65]
  Primary care visits | 891 [684 to 1097] | 1014 [745 to 1282]
  Other specialist visits | 257 [145 to 370] | 235.69 [159 to 313]
  Emergency department visits | 34 [-6 to 75] | 23 [-2 to 48]
  Inpatient admissions | 6495 [4565 to 8426] | 6140 [4160 to 8120]
  Indirect costs | 23 [13 to 33] | 14 [6 to 22]
  out-of-pocket costs | 114 [75 to 153] | 93 [50 to 136]
  Total costs | 7813 [5660 to 9966] | 7538 [5488 to 9588]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.955, t-test, 2 sided; Mean Difference (Final Values) = 275.00, 95% CI 2-sided [-3288 to 2739], Standard Error of Mean 1525

28. Secondary Outcome: Change From Baseline in Sleep Latency (Minutes)
Description: Sleep latency is the time it takes to fall asleep after turning the lights out.
Time Frame: Baseline to 6 months and 12 months
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
minutes
  6 month change | -14.06 (2.24) | -0.17 (2.30)
  12 month change | -10.86 (2.09) | -1.83 (2.19)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.0130, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

29. Secondary Outcome: Change in Sleep Latency
Description: Sleep latency is the amount of time it takes to fall asleep after turning off the lights.
Time Frame: Baseline to 3 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
minutes | -4.39 (43.97) | -2.11 (44.28)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.7496, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = -0.05

30. Secondary Outcome: Change in Sleep Related Impairment
Description: We used the 8-item PROMIS Sleep-Related Impairment questionnaire to measure self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep problems. The instrument uses a 7-day time frame and a 5-point rating scale that ranges from 1 ("Not at all") to 5 ("Very much"). The measure uses a T-score metric in which 50 is the mean of a relevant reference population (the general population) and 10 is the standard deviation (SD) of the population. Higher scores mean more sleep related impairment. To find the total raw score we summed the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40. We used the score conversion table to translate the total raw score into a T-score for each participant. The T-scores are interpreted as follows: Less than 55 = None to slight 55.0-59.9 = Mild 60.0-69.9 = Moderate 70 and over = Severe.
Time Frame: Baseline to 3 months
Population: Modified Intent to treat
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score | -8.56 (9.5) | -7.54 (11.4)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.3821, GLMM — [p-value comment as in outcome 2, analysis 1]; effect size = 0.06

31. Secondary Outcome: Change From Baseline in Sleep Related Impairment
Description: as for outcome 30
Time Frame: Baseline to 6 months and 12 months
Population: Modified intent to treat
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
Number analyzed (Participants) | 91 | 84
T-score
  6 month change | -10.23 (1.03) | -9.54 (1.08)
  12 month change | -10.74 (0.98) | -10.23 (1.05)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Heart Failure Self-Management Education; Test type: Superiority; p = 0.7204, Mixed Models Analysis — The p value is from the group X time interaction adjusted at 12 months based on the false discovery rate

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cognitive Behavioral Therapy | Heart Failure Self-Management Education
All-Cause Mortality (participants affected / at risk) | 0/91 | 8/84
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/84
Other Adverse Events (participants affected / at risk) | 0/91 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02660385/Prot_SAP_000.pdf